CLINICAL TRIAL: NCT04258826
Title: A Single-Dose Study Using Functional Magnetic Resonance Imaging to Evaluate the Effect of LY3154207 in Healthy Subjects
Brief Title: A Study to Evaluate LY3154207 on the Brain of Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17294; I7S-MC-HBEM (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02-15

CONDITIONS: Healthy
MeSH Terms: interventions — LY3154207

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3154207 (Experimental): LY3154207 administered orally in one of two study periods.
  Interventions: Drug: LY3154207
- Placebo (Placebo Comparator): Placebo administered orally in one of two study periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3154207 — LY3154207 administered orally.
  Arms: LY3154207
Drug: Placebo — Placebo administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about how LY3154207 affects the brain of healthy participants by using magnetic resonance imaging. The study will last up to about nine weeks for each participant and may include up to four visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

-Overtly healthy males and non-childbearing females, as determined through medical history and physical examination

Exclusion Criteria:

* Have known or ongoing psychiatric disorders
* Have contraindications to magnetic resonance imaging (MRI)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Intrinsic Functional Connectivity Among Resting-State Networks of the Brain | Day 1, Approximately Day 28
  Mean Connectivity and Mean Component Weight Between LY3154207 and Placebo in the Dorsal Attention Network (DAN), Frontoparietal Network (FPN), and Executive Control Network (ECN).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No